CLINICAL TRIAL: NCT01325324
Title: Comparison of Different Portable Tonometers (Icare Pro, TONO-Pen AVIA, Perkins Tonometer, PASCAL Hand Held Dynamic Contour Tonometer)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: portable-Tono-Study
Record Dates: First submitted 2011-03-14; First posted 2011-03-29 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Other): Study group
  Interventions: Device: measurement of intraocular pressure

INTERVENTIONS:
Device: measurement of intraocular pressure — Intraocular pressure will be measured with the following devices (each 2 times)at the first and only study visit
  Other Names: Icare Pro (Icare Finland Oy, Espoo, Finland); TONO-Pen AVIA (Reichert Terchnologies Inc., Depew, NY; USA; Perkins Tonometer (Haag-Streit AG, Könitz, Switzerland); PASCAL hand helt-Dynamic Contour Tonometer (Ziemer Ophthalmic Systems AG, Port, Switzerland)

SUMMARY:
In different cases intraocular pressure (IOP) have to measured in lying position. Therefore a lot of portable tonometers have been established. The Icare Pro is a new tonometer on the market that allows faster and more comfortable IOP-measurements. No local anesthesia is needed, what is a major advantage for the patients. In this study the investigators want to evaluate if IOP measurements with Icare Pro Tonometer are as reliable as they are with other established portable tonometers (Perkins, TONO-Pen and hand held-Dynamic Contour Tonometer).

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* healthy patients of at least 18 years of age or above

Exclusion criteria:

* diagnosis of glaucoma or other optic neuropathies
* corneal disorder that make IOP measurement impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | Study Visit 1
  the intraocular pressure will be measured at the first and only study visit (Visit 1, day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Funk, Prof. MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schweier C, Hanson JV, Funk J, Toteberg-Harms M. Repeatability of intraocular pressure measurements with Icare PRO rebound, Tono-Pen AVIA, and Goldmann tonometers in sitting and reclining positions. BMC Ophthalmol. 2013 Sep 5;13:44. doi: 10.1186/1471-2415-13-44. PMID 24006952